CLINICAL TRIAL: NCT07087730
Title: Improving Patient Mental Health With Psychotherapist Virtual Training: A Practice- Research Network Study
Brief Title: Improving Patient Mental Health With Psychotherapist Virtual Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: University of Toronto (Other); Sinai Health System (Other)
Responsible Party: Principal Investigator, Giorgio A. Tasca, Principal Investigator, Full Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 156261; 461713 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-04-23; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Mental Disorders
Keywords: Psychotherapists; Psychotherapy; Outcome Assessment, Healthcare; Cultural Diversity; Humans; Mental Disorders; Telemedicine
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: 3-arm, prospective, single blind randomized controlled trial with 2-1-1 allocation comparing (i) Virtual training, (ii) training as usual, (iii) no training.
Who Masked: Participant
Masking Description: Patients will be blind to therapist study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Training Program (Experimental): Asynchronous virtual training professional development program including consultation.
  Interventions: Behavioral: Virtual Training Program
- Training as Usual (Active Comparator): Synchronous virtual workshop professional development including consultation.
  Interventions: Behavioral: Training as Usual
- No Training (Active Comparator): No training, therapy as usual.
  Interventions: Behavioral: No Training

INTERVENTIONS:
Behavioral: Virtual Training Program — Therapists randomized to this condition will receive the professional development via an asynchronous virtual training course. The Virtual Training will include written material, videos, interactive learning activities, and a text-based discussion forum where therapists and faculty will be able to interact in relation to the given activities. Clinical scenario and simulation-based interactive learning will allow therapists to explore clinical situations, make decisions, and evaluate consequences of their actions in a safe environment. Therapists will complete 6 study-related therapy sessions with 3 new patients. After therapists receive the Virtual Training and after they enroll their first patient, therapists will attend bi-weekly 1-hour online consultation meetings that include up to 6 therapists at a time and led by two of the training faculty. Each therapist will attend 10 of these posttraining consultation sessions.
  Arms: Virtual Training Program
Behavioral: Training as Usual — Therapists randomized to this condition will receive the professional development training via a 3-day synchronous workshop delivered via video conference covering the same didactic content as the virtual training course. The workshop will include lectures, written material, videos, and live role play activities. Therapists will complete 6 study-related sessions with 3 new patients. After therapists receive the professional development through Training as Usual and after they enroll their first patient, therapists will attend bi-weekly 1-hour online consultation meetings that include up to 6 therapists at a time and led by two of the training faculty. Each therapist will attend 10 of these posttraining consultation sessions.
  Arms: Training as Usual
Behavioral: No Training — Therapists randomized to this control condition will provide psychotherapy via the study video conference platform to 3 new enrolled patients in their typical manner except that they and their patients will also complete the assessments necessary for the study. After study completion, the investigators will provide therapists in the control condition with access to virtual training.
  Arms: No Training

SUMMARY:
Several types of psychotherapy are equally effective to treat mental disorders. However, many patients remain symptomatic after treatment. The investigators demonstrated that a professional development training program to improve psychotherapists' skills at identifying and repairing therapeutic alliance tensions resulted in improved therapeutic alliance (an important therapeutic ingredient) and patient mental health outcomes. However, the investigators delivered this training program by conventional in-person workshops which limited access by psychotherapists living outside large urban centres. Further, post-study interviews with therapists suggested that cultural/diversity factors complicated the therapeutic alliance.

In the current study, the investigators will test the effectiveness and acceptability of a virtually-delivered training program to psychotherapists in North America to improve their capacity to identify and repair problems in the therapeutic alliance, including tensions related to patient diversity. The investigators will also examine how acceptable the virtually-delivered training is to psychotherapists and whether they would use such training in their practice. Participants in the study will be community-based licensed psychotherapists and their patients engaging in therapy in North America. Patient mental health outcomes, therapeutic alliance, and diversity issues will be assessed by comparing outcome measures between three groups: 1) therapists complete a self-paced virtual course + consultation, 2) therapists complete synchronous workshop + consultation, 3) control: therapists do not complete training.

The team of investigators developed Canada's largest psychotherapy practice-research network and has expertise in clinical trials, diversity, and education research of virtual training. State of the art training is often out of the reach of therapists who live outside of urban centres, and the effectiveness and acceptability of providing training virtually is not well-studied in mental health care. This study will improve psychotherapists' effectiveness at managing the therapeutic alliance and issues related to diversity, and will improve patient mental health outcomes thus promising to reduce the burden of mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Therapist participants: The investigators will recruit mental health professionals who deliver psychotherapy in North American community settings; inclusion criteria: therapists are in good standing with their provincial or state regulatory college, their scope of practice includes individual psychotherapy for adults in North America; they are able to accept a minimum of 3 new participating patients into their current practice to conduct 6 consecutive therapy sessions via a secure, PHIPA compliant virtual meeting platform.
* Patient Participants: Adults (> 18 years) residing in Canada or the United States who want to engage in therapy with a study therapist or who have recently sought services from a study therapist; inclusion criteria: have participated in fewer than 3 sessions with their study therapist and anticipate being able to see their study therapist for 6 sessions over the next 6 months.

Exclusion Criteria:

* Therapist participants: The investigators will exclude therapists who are employed by an organization if the investigators cannot obtain organizational approval from their employer or coordinate data collection from an alternate virtual platform in instances where the employing organization does not permit the use of the study platform. Therapists will also be excluded if they have completed professional development workshop after 2017 with PPRNet.
* Patient participants: The investigators will exclude patients if they: (a) have a psychotic or neurocognitive disorder that may preclude engagement in psychotherapy, (b) are in concurrent psychological treatment with another practitioner, (c) are at high risk of suicide or suicidal behaviors as assessed by their therapist (e.g., suicide attempt or hospitalization for suicidal behaviors in the past 6 months), or (d) for whom the therapist judge that approaching them with information about the study will be harmful.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 489 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Working Alliance Inventory (WAI) therapist or patient short form | Patients and therapists will complete it after each of 6 consecutive study psychotherapy session (frequency will range from once a week to once a month depending on the client's typical session interval).
  12-item self-report measure used to assess the therapeutic alliance by either therapist or client. Yields scores on three subscales: task, bond, and goal. Min subscale score is 12, max score is 84 with higher scores indicate greater alliance.
Ruptures Resolution Rating System (3RS) | Sessions will be coded by trained raters after all session recordings have been collected.
  Observer-based coding system for identifying therapeutic alliance ruptures and resolutions.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Patients will complete it before starting study psychotherapy sessions, after completing all study sessions (6 weeks to 6 months depending on the client's typical session interval), and at 3-month follow-up.
  Self-report measure used to assess depressive symptoms. Min score is 0; max score is 27 with higher scores indicating greater severity of depressive symptoms.
Generalized Anxiety Disorder questionnaire (GAD-7) | Patients will complete it before starting study psychotherapy sessions, after completing all study sessions (6 weeks to 6 months depending on the client's typical session interval), and at 3-month follow-up.
  Self-report measure used to assess anxiety symptoms. Min score is 0; max score is 21 with higher scores indicating higher levels of anxiety symptoms.
Inventory of Interpersonal Problems (IIP-32) | Patients will complete it before starting study psychotherapy sessions (6 weeks to 6 months depending on the client's typical session interval), after completing all study sessions, and at 3-month follow-up.
  Self-report measure used to assess interpersonal problems. This 32-item measure yields 8 subscales with a min score of 0 and a max score of 15 per scale with higher scores indicating greater interpersonal problems.
Defense Mechanism Rating Scales (DMRS-SR-30) | Patients will complete it before starting study psychotherapy sessions, after completing all study sessions (6 weeks to 6 months depending on the client's typical session interval), and at 3-month follow-up.
  Self-report measure used to assess defense mechanisms. Total score can range from 0 to 120 with low scores indicate low adaptive functioning and higher scores indicate better adaptive functioning.
Experiences in Close Relationships (ECR-12) | Patients will complete it before starting study psychotherapy sessions and 3 months after completing therapy sessions. Therapists will completed it before receiving training.
  Self-report measure used to assess two dimensions of attachment: attachment avoidance and anxiety. Scores on each scale can range from 6 to 42 with high scores indicating greater attachment avoidance or anxiety.
Certainty About Mental States Questionnaire (CAMSQ) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess a person's perceived capacity to understand oneself and others' mental states. Mean scores of subscales can range from 1 to 7 with higher mean scores indicating higher mentalization.
Multidimensional scale of perceived social support (MSPSS) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess perceived adequacy of support from family, friends, and significant others. The mean score on each subscale can range from 1 to 7 with higher scores indicating greater social support.
Rosenberg Self-Esteem Scale (RSES) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess self-esteem. Total score can range from 0 to 30 with higher scores indicating higher self esteem.
Epistemic Trust, Mistrust, and Credulity Scale (ETMCQ) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess epistemic trust on three subscales: trust, mistrust, and credulity. Mean scores on each subscale ranges from 1 to 35 with higher scores indicating greater trust.
Outcome Rating Scale (ORS) | Patients and therapists will complete it after each of 6 consecutive study psychotherapy session (frequency will range from once a week to once a month depending on the client's typical session interval).
  4-item visual analogue scale used to assess global functioning for the previous week by indication their position on a rating line on 4 scales: personal wellbeing, family/close relationships, work/school/friendships; overall. Scores can be examined for each item that can create a total score for all items that can range between 0 to 40. Higher scores indicate higher functioning.
Schwartz Outcome Scale (SOS-10). | Patients will complete it before starting study psychotherapy sessions, after each study-related therapy session (over 6 weeks to 6 month period), and at 3-month follow-up; therapists will complete it after each study session (6 weeks to 6 months).
  Self-report measure used to assess well-being. A total score across items can range from 0 to 60 with higher scores representing greater psychological well-being and lower scores indicating emotional distress and poorer psychological health.
Multitheoretical List of Therapeutic Interventions (MULTI-30) | Therapists and patients will complete respective versions of the measure after completing all study therapy sessions (6 weeks to 6 months after the first study session depending on the frequency of study session).
  Self-report measure used to assess therapeutic interventions used in psychotherapy sessions. Weighted mean scores on 8 intervention subscales are calculated with a range of 1 to 5. Higher scores indicate intervention approaches that are very typical with lower scores indicating less typical.
Real Relationship Inventory (RRI) | Therapists and patients will complete respective versions of the measure after completing all study therapy sessions.
  Self-report measure used to assess the therapeutic relationship. Two subscales, realism and genuineness combined to generate a total score. Total scores range from 24 to 120 with higher scores indicating stronger relationship.
Patient drop-out | Patient drop-out will be monitored throughout the study.
  Unilateral withdrawal from treatment by a patient at any time during the study will indicate a negative outcome. The investigators will monitor whether drop out occurred early (<5 sessions) or late (>5 sessions).
Certainty About Mental States Questionnaire (CAMSQ) | Therapists will complete the measure before and after receiving training.
  Self-report measure used to assess a person's perceived capacity to understand oneself and others' mental states. Mean scores of subscales can range from 1 to 7 with higher mean scores indicating higher mentalization.
Trauma-informed Care Provider Survey (TICPS) | Therapists will complete the measure before and after receiving training.
  Self-report measure used to assess healthcare providers' knowledge, opinions, and competence related to trauma-informed care. Total score subscales are as follows: knowledge, can range from 13 - 52; opinions toward trauma-informed, can range from 7-28; competence can range from 0-24. with higher scores indicating more knowledge, opinions favourable to trauma-informed care, and competence.
Gay Affirmative Practice Scale (GAP) | Therapists will complete the measure before and after receiving training.
  Self-report measure used to assess practitioners' engagement with gay-affirmative practices on two subscales; beliefs and behaviour. Scores on the each subscale can range from 15 to 75 with higher total across subscales reflecting more affirmative practice with gay and lesbian clients.
Multicultural Counseling Self-Efficacy Scale | Therapists will complete the measure before and after receiving training.
  Self-report measure used to assess therapists' perceived ability to counsel culturally diverse patients. A mean total scale score is calculated, ranging from 0 to 9, with higher scores indicating stronger multicultural counseling capabilities.
Psychologist and Counselor Self-Efficacy Scale (CASES) | Therapists will complete the measure before and after receiving training.
  Self-report measure used to assess therapists' professional self-efficacy on three domains: basic helping skills, session tasks, and challenging counseling situations and presenting issues with scores ranging from 0 to 135 with greater scores indicating greater perceived efficiency.
Adverse Childhood Experiences - Philadelphia version (Philly-ACES) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess the number of adverse childhood experiences across 14 categories. The number of adverse experiences across categories is summed and participants are given one of the following scores: 0, 1-2, or 3+ Adverse Childhood Experiences.
Trauma Symptom Discrimination Scale (TSDS) | Patients will complete it before starting study psychotherapy sessions.
  Self-report measure used to assess distress and anxiety symptoms due to the experience of discrimination. A total score is calculated by adding up the scores from all items and can range from 21 to 84 with higher scores indicating higher distress due to experiences of discrimination.

OTHER OUTCOMES:
Cultural Humility Scale (CHS) | Patients will complete the measure after completing all study therapy sessions.
  Patient-rated measure of a therapist's cultural humility. A total score is calculated and ranges from 12 to 60. Higher total scores reflect greater levels of cultural humility.
Sexist Microaggression Scale (MAWS) | Patients who self-identify as women will complete it after each study psychotherapy session (over 6 weeks to 6 months depending on the frequency of sessions).
  Self-report measure used to assess women's experience of microaggressions during psychotherapy sessions. Total score can range from 7 to 35 with higher scores representing greater experiences of microaggressions from the therapists.
Racial Microaggressions in Counseling Scale (RMSC) | Patients who self-identify with a marginalized race will complete it after each study psychotherapy session. Sessions will occur over a 6 week to 6 month period depending on the frequency of sessions.
  Self-report measure used to assess racialized patients' experience of microaggressions during psychotherapy sessions. An average total score is calculated ranging from 1 to 3 with higher scores indicate greater frequency and impact of microaggressions.
Sexual Orientation Microaggressions in Psychotherapy Scale (SOMPS) | Patients who self-identify as lesbian, gay, bisexual, or queer will complete it after each study psychotherapy session (sessions will occur over a 6 week to 6 month period depending on the frequency of sessions).
  Self-report measure used to assess lesbian, gay, bisexual, or queer patients' experience of microaggressions during psychotherapy sessions. An average total score is calculated ranging from 1 to 3 with higher scores indicate greater frequency and impact of microaggressions.
Gender Identity Microaggressions scale (GIMS) | Patients who self-identify as trans or non-binary will complete it after each study psychotherapy session. Psychotherapy sessions will occur over 6 weeks to 6 months depending on the frequency of sessions.
  Self-report measure used to assess trans or non-binary patients' experience of microaggressions during psychotherapy sessions. Total scores can range from 8 to 40 with higher scores indicating greater experiences of microaggressions.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio A Tasca, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: recruitment site — https://researchpprnet.ca/